CLINICAL TRIAL: NCT03216434
Title: Striatal Dopamine Transporter Density in Post-Traumatic Stress Disorder (PTSD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Principal Investigator, Pam Dewey, research clinician, St. Joseph's Hospital and Medical Center, Phoenix
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PHXB-17-0104-71-21
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Post-traumatic Stress Disorder
Keywords: post-traumatic stress disorder; dopamine; biomarker
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PTSD Diagnosed (Experimental): Veterans exposed to combat and diagnosed with PTSD. MRI using DaTscan.
  Interventions: Diagnostic Test: MRI using DaTscan
- Designated Combat-Experienced Controls (Experimental): Veterans exposed to combat, but never diagnosed with PTSD. MRI using DaTscan.
  Interventions: Diagnostic Test: MRI using DaTscan

INTERVENTIONS:
Diagnostic Test: MRI using DaTscan — A standard, non-contrast-enhanced structural/anatomic brain MRI will be performed. It will be used to exclude potential subjects and controls with significant and potentially confounding structural/anatomic findings. It will also be used as an "anatomic overlay" with the functional DaTscan image to aid in anatomic/physiologic correlation. At the same imaging session, a brief functional MRI (not requiring the subject to perform any tasks) will also be performed.

SUMMARY:
This research study is being done to try to find a way to accurately diagnose post-traumatic stress syndrome (PTSD) in combat veterans.Diagnostic biomarkers have made invaluable contributions to the diagnosis and treatment monitoring of many diseases and disorders. Unfortunately, PTSD currently lacks a reliable and compelling clinically-relevant biomarker. The absence of a viable biomarker impairs efficient and confident diagnosis of PTSD, with diminished effective care options often resulting.

DETAILED DESCRIPTION:
The possibility of developing PTSD exists when a person is exposed to death, threatened death, or actual or threatened serious injury either by direct exposure, witnessing the trauma, or learning that a close friend was exposed to this type of trauma. Rates of PTSD in military personnel returning from armed conflicts may be greater than 30%. The diagnosis of PTSD is based on a psychiatrist's or psychologist's assessment of the symptoms reported by the veteran and others, such as family or friends.The veteran with PTSD may struggle with thoughts and feelings that "don't make sense" or he or she believes are just not "warrior-like". The veteran eventually sees a mental health professional but may downplay the symptoms and fail to be correctly diagnosed. This places these men and women at risk for suicide. Dopamine is a substance found in our brains that has a role in regulating fear and stress as well as other emotional responses. There have been studies that have shown a protein in blood called dopamine transporter (DAT) moves dopamine from one place to another in our brain. Studies have shown that the level of DAT present has a role in PTSD. In this research, the researchers will evaluate the usefulness of a type of radioactive drug (DaTscan) which attaches to DAT and then allows the researchers to take pictures of the brain using a camera called a gamma camera. This will produce images called single photon emission computed tomography (SPECT). The researchers are looking for a difference in these pictures in those with PTSD and veterans without PTSD, and hope this can be used to help diagnose PTSD in the future.The brain MRI is done to make sure there is not anything abnormal in the structure of the brain that could interfere with the DaTScan pictures and to accurately locate specific regions of the brain where the DaTScan pictures are especially important. The MRI will also be used to look at natural nerve connections in the brain using functional MRI or fMRI. The researchers will use fMRI to look for possible connection differences in brains of people with PTSD and without PTSD. The DaTscan requires a drug, called a radiotracer given through an intravenous (IV) catheter. This drug is radioactive and a small amount of it will be absorbed by the thyroid gland, so Lugol's solution will be used to block uptake into the thyroid. The length of time to complete the entire DaTscan process is approximately 5 ½ hours. This includes time to receive the drug, then a 3 hour break followed by about 45 minutes to take the pictures. The tracer will collect in part of the brain and give off radiation (gamma rays). A gamma camera will produce pictures of the brain.The MRI process will take approximately 1 hour, including a questionnaire about metal or implants in the subject's body. Brain scanning will last for about 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Diagnosed with PTSD (n=25) or designated combat-experienced controls (n=25)

Exclusion Criteria:

* Head trauma resulting in loss of consciousness
* Co-morbid DSM IV Axis I psychiatric disorder
* hyper- or hypo-thyroidism, neurological motor deficits (e.g. Parkinsonism, tremor)

Ages: 22 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
DaTscan intensity | within 30 days of MRI
  Visually recognizable increases in striatal DaTscan intensity in PTSD patients.
Quantifiable differences | within 30 days of MRI
  Quantifiable differences in global and regional DAT density in PTSD patients and combat-experienced controls.

SECONDARY OUTCOMES:
Striatal correlations | within 60 days of entry into study
  Global and regional striatal correlations of DAT density with elements of the psychological/psychiatric evaluation (i.e. psychological/ psychiatric symptoms). For example, the researchers will examine the correlation of DAT density with sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Frank V Schraml, MD, Principal Investigator — St. Joseph's Hospital and Medical Center, Phoenix

IPD SHARING:
Plan to Share IPD: No